CLINICAL TRIAL: NCT06011304
Title: A Phase III, Open-Label, Multi-center Clinical Study to Assess the Diagnostic Performance and Safety of 18F-Florastamin PET/CT Imaging in Patients With at Least Intermediate Risk Prostate Cancer
Brief Title: Study of 18F-Florastamin PET/CT Imaging in Patients With at Least Intermediate Risk Prostate Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: HTA Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BJK-ZX-STM-2202-GK
Record Dates: First submitted 2023-08-21; First posted 2023-08-25 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-Florastamin Injection (Experimental)
  Interventions: Drug: [18F]Florastamin Injection

INTERVENTIONS:
Drug: [18F]Florastamin Injection — The subjects who participate in phase 3 study will be intravenously injected with [18F]Florastamin Injection and undergo PET/CT scan at 110 min after the injection.
  Subjects who participate in pilot study will be intravenously injected with [18F]Florastamin Injection and undergo PET/CT scan at 5 min, 30 min, 60 min, 110 min, 160 min after the injection.

SUMMARY:
In this study, 18F-Florastamin PET/CT will be performed in patients with at least intermediate risk prostate cancer, to assess the diagnostic performance and safety of 18F-Florastamin PET/CT imaging.

This study will first carry out the pilot study (including pharmacokinetics and radiation dosimetry).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects fully understood the content, process, and potential risks of the study and voluntarily signed an informed consent form (ICF).
2. Male subjects aged 18 or older.
3. Subjects with histopathological diagnosis of prostate adenocarcinoma.
4. According to clinical judgment, radical prostatectomy and pelvic lymph node dissection (which can include patients with localized, regional lymph node metastasis or oligometastatic prostate cancer) are planned, and there is no surgical contraindication.
5. If it is localized prostate cancer, according to the Prostate Cancer Diagnosis and Treatment Guidelines of 2021 Chinese Society of Clinical Oncology, it is necessary to meet any of the following criteria:

   Intermediate Risk: Has at least one intermediate risk factor: T2b-T2c; Gleason pattern 2 or 3; PSA 10-20 ng/mL, and does not include feature of high-risk or very-high-risk groups.

   High Risk: Has no very-high-risk features and has at least one high-risk feature: T3a; Gleason Grade Group 4 or 5; PSA >20 ng/mL.

   Very High Risk: Has at least one of the following: T3b-T4; Primary Gleason pattern 5; More than 4 punctures with Gleason Grade Group 4 or 5.
6. ECOG score 0 or 1.
7. Subjects who meet the following conditions in hematology, renal function, and liver function:

   * Platelet count>100 * 10^9/L
   * Urea nitrogen and creatinine<1.5 times upper limits of normal
   * AST and ALT<2.5 times upper limits of normal.
8. Expected survival time ≥ 6 months.
9. Subjects and their partners must use effective contraceptive measurements and avoid sperm donation from the date of signing ICF to 3 months after administration.

Exclusion Criteria:

1. Subjects who have participated in other interventional clinical trials before signing ICF and were within the 5 half-lives of the investigational drug, or who are currently participating in other interventional clinical trials or have participated in clinical trials of radioactive drugs within 1 year before signing ICF and have been discontinued for less than 3 months until the signing date of ICF.
2. Intravenous injection of iodinated contrast medium within 24 hours, or any high-density oral contrast medium (Such as barium sulfate. Oral water contrast is acceptable, such as compound meglumine diatrizoate oral liquid) within 5 days, prior to study drug administration.
3. Subjects administered any high energy (>300 KeV) gamma-emitting radioisotope within five physical half-lives prior to study drug administration.
4. Patients with prior androgen deprivation therapy or any other neoadjuvant agent.
5. The investigator determines that there are any medical diseases or other conditions that affect the safety or compliance of the subjects.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Specificity | Within 28 days following 18F-Florastamin PET/CT
  The specificity of 18F-Florastamin PET/CT in patients with negative pelvic lymph node metastasis compared with the histopathology.
  The subjects underwent RP (radical prostatectomy) with PLND (pelvic lymph node dissection) within 28 days after the administration of 18F-Florastamin Injection. The histopathology results of the pelvic lymph node tissue collected from the subjects will be used as the standard of truth for this study.

SECONDARY OUTCOMES:
Sensitivity | Within 28 days following 18F-Florastamin PET/CT
  The sensitivity of 18F-Florastamin PET/CT in patients with positive pelvic lymph node metastasis compared with the histopathology.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, China